CLINICAL TRIAL: NCT00481806
Title: Thrombin Dysregulation Leads to Early Saphenous Vein Graft Failure
Brief Title: Evaluating the Role of Thrombin in Saphenous Vein Graft Failure After Heart Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: University of Maryland, Baltimore County (Other)
Responsible Party: Principal Investigator, Robert Poston, Chief, Division of Cardiothoracic Surgery, University of Arizona
Other Study IDs: 479; R01HL084080-01A1 (NIH)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Bypass; Thrombosis
Keywords: Virchow's Triad; Thrombin; Graft Failure
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and vein samples

SUMMARY:
Heart bypass surgery, also known as coronary artery bypass graft (CABG) surgery, creates a detour around the blocked part of a heart artery to restore blood supply to the heart muscle. The saphenous vein, located along the inside of the leg, is commonly used to create the bypass in a CABG surgery. An abnormal increase in the blood clotting protein thrombin may cause the saphenous vein graft to close up and eventually fail. This study will evaluate the relationship between thrombin levels and saphenous vein graft failures in people undergoing a CABG procedure.

DETAILED DESCRIPTION:
The saphenous vein, which runs from the ankle to the groin along the inside of the leg, is commonly used as a graft for people undergoing a CABG surgery. The vein is removed from the leg and reattached to the heart to create a detour around the blocked part of a coronary artery. Following this procedure, many people are prescribed aspirin as a way to increase the chance that the graft procedure will be successful. However, saphenous vein graft failure may still occur in some people, indicating a need to understand why this happens and who might be at risk for graft failure. Thrombin, a protein involved in the blood clotting process, is somehow related to aspirin resistance, abnormalities in blood flow, and cell disruption within the saphenous vein, all factors thought to increase the risk of graft failure. The purpose of this study is to evaluate the likelihood that a burst in thrombin contributes to graft failure in people who have recently undergone a CABG procedure using the saphenous vein.

This study will enroll individuals undergoing CABG surgery at the University of Maryland. Prior to and immediately following surgery, an incision will be made in the skin and the time required for the blood to form a clot will be determined. During surgery, participants' blood vessels will be examined using imaging and cell analysis techniques. Blood collection will occur before surgery, immediately after surgery, and on Days 1, 3, and 30 following surgery. A portion of blood will be frozen for future analysis. An x-ray of the saphenous vein will be performed on Day 5 and again at a follow-up visit 6 to 12 months following surgery. Kidney function will be measured at both of these visits prior to the x-ray procedure. At the second visit, health and mental status questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for CABG surgery at University of Arizona University Medical Center (UMC)
* For females, willing to use a reliable form of birth control for the duration of the study

Exclusion Criteria:

* Non-dermatologic allergy to intravenous (IV) radiographic contrast
* Creatinine levels greater than 2.0 mg/dL
* Pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients between the the age of 18-90 years belonging to all races will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2007-02; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Amplifying the severity of all three risk factors of Virchow's triad is expected to lead to a synergistic increase in regional thrombin formation | Measured at 5 years
Pressure distention is the main stimulus that creates a loss of thrombin control within the SVG | Measured at 5 years
Accurate tests of graft quality will be developed that provide rapid results for ready translation into clinical applications | Measured at 5 years
Aprotinin or bivalirudin will effectively suppress thrombin generation and its effects within the highest risk grafts | Measured at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Poston, MD, Principal Investigator — University of Arizona, Tucson
Locations (1):
- University of Arizona College of Medicine, Tucson, Arizona, United States

REFERENCES:
- [Derived] Desai P, Kiani S, Thiruvanthan N, Henkin S, Kurian D, Ziu P, Brown A, Patel N, Poston R. Impact of the learning curve for endoscopic vein harvest on conduit quality and early graft patency. Ann Thorac Surg. 2011 May;91(5):1385-91; discussion 1391-2. doi: 10.1016/j.athoracsur.2011.01.079. PMID 21524447
- [Derived] Poston RS, Tran R, Collins M, Reynolds M, Connerney I, Reicher B, Zimrin D, Griffith BP, Bartlett ST. Comparison of economic and patient outcomes with minimally invasive versus traditional off-pump coronary artery bypass grafting techniques. Ann Surg. 2008 Oct;248(4):638-46. doi: 10.1097/SLA.0b013e31818a15b5. PMID 18936577